CLINICAL TRIAL: NCT04588155
Title: Temporal and Kinematic Analysis of Timed Up and Go Test in Chronic Low Back Pain
Brief Title: Temporal and Kinematic Analysis of Timed Up and Go Test in Chronic Low Back Pain Patients
Status: Completed | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Principal Investigator, Riccardo Buraschi, Principal Investigator, Fondazione Don Carlo Gnocchi Onlus
Other Study IDs: TUGLBP_FDG
Record Dates: First submitted 2020-09-17; First posted 2020-10-19 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Chronic Low-back Pain
Keywords: Chronic Low-back Pain; Functional assessment; Time Up and Go Test; Inertial measurement unit

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic Low-Back Pain: Subjects diagnosed with Chronic Low-Back Pain in rehabilitation program: functional assessment (with temporal and kinematic analysis) and clinical assessment.
  Interventions: Device: Functional assessment; Other: Clinical assessment
- Healthy: Healthy subjects: functional assessment (with temporal and kinematic analysis)
  Interventions: Device: Functional assessment

INTERVENTIONS:
Device: Functional assessment — Timed Up and Go Test administration with application of Inertial Measurement Unit for a temporal and kinematic assessment of movement performed during test esecution
Other: Clinical assessment — Roland Morris Disability Questionnaire (RMDQ) to assess the level of functional impairment and disability in the activity of daily living
  Numerical Pain Rating System (NPRS) administration to quantify level of pain experienced just before the TUG test execution
  Groups: Chronic Low-Back Pain

SUMMARY:
Kinematic and temporal analysis of the movement helps researchers and clinicians to better understand the way humans move and interact within the environment in which they live, better describe the alterations coming from impairments, and finally allow to better tailor interventions for patients. In this perspective, motion analysis has become, in the last 30 years, a remarkable and important field of research. Even if movement assessment should be a cornerstone for definition and modulation of rehabilitation interventions, there are still few motion analysis devices that are able to influence the clinical decision process; motion analysis labs are among those, but their use is unfortunately limited due to the costs of instruments and analysis. Other small unobtrusive wearable devices, easier to use and cost-effective, have been developed, like Inertial measurement units (IMU), composed by accelerometers and gyroscopes. They could therefore represent an incentive for a more widespread use of motion analysis within daily clinical activity in Rehabilitaion.

Timed Up and Go Test (TUG) is a simple, widely used, functional test which involves standing up from a chair, walking three meters, turning, and going back to sit. It is used to evaluate movement, mobility, dynamic and static balance in people with musculoskeletal impairment, neurological diseases, aging related conditions, and the quality of life in people with low back pain. The only and easy outcome considered is the time to completion. Nevertheless, the application of an IMU to a subject performing TUG can provide other objective, quantitative data, like temporal and kinematic parameters of the whole test and its sub-phases. The instrumented TUG (iTUG) has already been applied, mainly in the neurorehabilitation field, in particular for Parkinson's disease and for post-stroke impairments.

cLBP is one of the most burdensome health problem worldwide. cLBP has been considered a bio-psycho-social disease, characterized by pain in the lumbar region, functional impairments, and condition-related disability. Despite the obvious motor problems affecting people with cLBP, to the best of our knowledge, chronic low back pain (cLBP) has not yet been explored using iTUG.

The aim of study is to analyse temporal and kinematic parameters of cLBP subjects compared to BMI and age-matched healthy subjects, through iTUG and to explore the correlations of those parameters with pain and disability.

ELIGIBILITY:
Inclusion Criteria (for Chronic Low Back Pain population):

* Pain from at least 3 months
* Numerical Pain Rating Scale (NPRS) ≥ 4

Exclusion Criteria (for Chronic Low Back Pain population):

* History of neurological impairment or disease,
* Other orthopaedic impairment within the past 6 months or surgery in the previous 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Population of Chronic Low Back Pain subjects participating to an outpatient rehabilitation program; Population of healthy subjects, age and BMI-matched with the Low Back Pian sample.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Temporal parameters of movement | through study completion, an average of 2 month
  Temporal analysis of TUG performance
Kinematic parameters of movement | through study completion, an average of 2 month
  Kinematic analysis of TUG performance

SECONDARY OUTCOMES:
Roland Morris Disability Questionnaire | through study completion, an average of 2 month
  Questionnaire that assess levels of impairment and disability coming from low back pain The score can range from 0 (no disability) to 24 (severe disability).
Numerical Pain Rating Scale | through study completion, an average of 2 month
  Scale for pain assessment: the minimum value "0" and maximum values "10", where higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Don Carlo Gnocchi Onlus - Centro Ettore Spalenza, Rovato, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Buraschi R, Pollet J, Villafane JH, Piovanelli B, Negrini S. Temporal and kinematic analyses of timed up and go test in chronic low back pain patients. Gait Posture. 2022 Jul;96:137-142. doi: 10.1016/j.gaitpost.2022.05.027. Epub 2022 May 26. PMID 35635989